CLINICAL TRIAL: NCT01695876
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), Food Effect of AMG 357 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110246; Inflammation (Other: Amgen)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-01

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- AMG 357 (Experimental): AMG 357 is a small molecule for treatment of inflammatory disease
  Interventions: Drug: AMG 357
- Placebo (Placebo Comparator): Matching placebo to AMG 357 containing no active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 357 — Oral administration available in varying dose strength.
  Arms: AMG 357
Drug: Placebo — Matching placebo to AMG 357 containing no active drug
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, PK, PD, and food effect of AMG 357 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult subjects between 25 and 55 years old
* Body mass index (BMI) between 18 and 32 kg/m2
* Normal or clinically acceptable physical examination, clinical laboratory values, and ECG
* Additional inclusion criteria apply

Exclusion Criteria:

* Any history or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety.
* Additional exclusion criteria apply

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 35 days
  Examine the number of adverse events per subject, and subject incidence of clinically significant changes in physical examinations, vital signs, laboratory safety tests and electrocardiograms, after single and multiple dose administration of AMG 357 in healthy subjects.

SECONDARY OUTCOMES:
Pharmacodynamics | up to 35 days
  Measure the area under the plasma concentration curve versus time of AMG 357 after single and multiple dose administration in healthy subjects
Effect of Food on AMG 357 | up to 11 days
  To assess the effect of food on the PK parameters of AMG 357

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- New Zealand (3):
  - Research Site, Christchurch
  - Christchurch
  - Research Site, Grafton, Auckland

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com